CLINICAL TRIAL: NCT04531293
Title: Mono-centred, Controlled Cross-over Study Comparing Pressure Based, and Dilution Based Total Lung Capacity Measurements in COPD Patients and Healthy Subjects Using Two Commercially Available Devices for Lung Function Diagnostics
Brief Title: Comparing Pressure Based and Dilution Based Total Lung Capacity Measurements in COPD Patients for Lung Function Diagnostics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ndd Medizintechnik AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EOP17
Record Dates: First submitted 2020-08-18; First posted 2020-08-28 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: COPD
Keywords: COPD; DLCO; spirometry; alveolar volume; body plethysmography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total-breath method followed by standard method (Other): Total Lung Capacity (TLC) measurement performed on device EasyOne Pro (TM) according to total-breath method followed by TLC measurement performed on device MasterScreen (TM) according to standard method.
  Interventions: Device: Respiratory Analysis System
- Standard method followed by total breath method (Other): Total Lung Capacity (TLC) measurement performed on device Masterscreen (TM) according to standard method followed by TLC measurement performed on device EasyOne Pro (TM) according to total-breath method.
  Interventions: Device: Respiratory Analysis System

INTERVENTIONS:
Device: Respiratory Analysis System — Measurement of total lung capacity using total-breath method
  Other Names: EasyOne Pro (TM) by ndd Medizintechnik AG
Device: Respiratory Analysis System — Measurement of total lung capacity using standard method
  Other Names: Masterscreen (TM) by Vyaire

SUMMARY:
Total Lung Capacity (TLC) of the lungs can be determined using a pressure based method (i.e. by body plethysmography) or it can be determined using a dilution based method (i.e. by single breath dilution during a CO diffusing capacity test). The results of the two methods differ, especially in patients with higher grades of COPD. The study investigates an improved analysis for the determination of TLC using the dilution method; this method has been suggested in the new ATS/ERS DLCO (diffusion capacity of lung for carbon monoxide) standard published in 2017. This study is based on approx. 120 participants. So far, there has not been a study using commercially available equipment.

Spirometry, lung volume measurement by body plethysmography and DLCO measurements will be performed on reference device (Masterscreen Body/Diff, Vyaire, USA), Spirometry and DLCO will also be performed on the device under test (EasyOne Pro LAB, ndd Medizintechnik AG, Switzerland) in a crossover design. Both devices are CE marked and FDA approved. The tests performed on both devices are standardized tests performed routinely with patients.

ELIGIBILITY:
Inclusion Criteria:

3 groups

* Healthy subjects, FEV1/FEV1(pred) > 80%
* COPD GOLD classification 1 or 2, FEV1/FEV1(pred) ≥ 50%
* COPD GOLD classification 3 or 4, FEV1/FEV1(pred) < 50%

Exclusion Criteria:

* Smoked during 2 hours prior to measurements

Additional exclusion criteria for healthy subjects:

* BMI > 30
* Any relevant concomitant diseases (investigators decision)
* Any relevant concomitant medication (investigators decision)
* FEV1/FEV1(pred) <= 80%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Comparison of Total Lung Capacity (TLC) measurement using total-breath method and standard method | single measurement on day 1
  Difference in Total Lung Capacity (TLC) using total-breath method (according to ATS/ERS standard 2017, EasyOne Pro) and TLC using normal dilution method (according to ATS/ERS standard 2005, EasyOne Pro) in relation to TLC using body plethysmography (Vyaire).

SECONDARY OUTCOMES:
Dependency between primary outcome and COPD disease severity | single measurement on day 1
  Correlation between ( TLC(dilution, total-breath, EasyOne Pro) - TLC(dilution, standard 2005, EasyOne Pro) ) / TLC(body, Vyaire) and FEV1(EasyOne Pro) / FEV1(predicted)
Device comparison using the same method for both devices. | single measurement on day 1
  Total Lung Capacity (TLC) (dilution, standard 2005, EasyOne Pro) / TLC(dilution, standard, Vyaire). Determines accuracy and comparability of both devices in measurement of TLC.

CONTACTS AND LOCATIONS:
Locations (1):
- LungenZentrum Hirslanden, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorres RA, Buess C, Piecyk A, Thompson B, Stanojevic S, Magnussen H. The total-breath method yields higher values of DLCO and TLC than the conventional method. BMC Pulm Med. 2024 Mar 13;24(1):127. doi: 10.1186/s12890-024-02932-y. PMID 38475751